CLINICAL TRIAL: NCT02662790
Title: Effects of Antenatal Dexamethasone Administration on Fetal and Uteroplacental Doppler Waveforms in Women at Risk for Preterm Birth
Brief Title: Dexamethasone on Fetal and Uteroplacental Doppler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEXA
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

ARMS (1):
- Preterm (Experimental)
  Interventions: Other: Doppler

INTERVENTIONS:
Other: Doppler

SUMMARY:
The current study aims to investigate the effects of dexamethasone exerted on fetal and uteroplacental circulation as measured by Doppler ultrasonography in pregnancies at risk for preterm birth after 24 hours of its administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk of preterm labor to be included were those with preterm uterine contractions, placenta previa, and mild preeclampsia

Exclusion Criteria:

* Patients who were actively in labor, presented with premature rupture of membranes, intrauterine growth restriction (IUGR), those who had received corticosteroids in their pregnancies and/or fetuses with suspected structural abnormalities

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
mean of Doppler Resistance index (RI) | 24 hours

SECONDARY OUTCOMES:
mean of Doppler Pulsatility index (PI) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt